CLINICAL TRIAL: NCT01866085
Title: Randomised Clinical Trial to Evaluate Efficacy of AdVance® vs ARGUS® Sling Procedure in Male With Post Prostatectomy Stress Urinary Incontinence
Brief Title: AdVance® vs ARGUS® Sling Procedure in Male With Post Prostatectomy Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish General Hospital (Other)
Collaborators: Center Hospitalier de Fleurimont,Sherbrooke University (Unknown); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jacques Corcos, MD. Professor of Urology, McGill University, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-013; 12-013 (Other: Research Ethics Board,JGH)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; post prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AdVance (Active Comparator): sling procedure
  Interventions: Procedure: AdVance® sling procedure
- ARGUS (Active Comparator): sling procedure
  Interventions: Procedure: ARGUS Sling procedure

INTERVENTIONS:
Procedure: AdVance® sling procedure
  Arms: AdVance
Procedure: ARGUS Sling procedure
  Arms: ARGUS

SUMMARY:
The study is designed to assess efficacy and subject satisfaction of two sling devices: Advance and Argus, in male patients with stress urinary incontinence after prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male
* The subject is at least 18 years of age
* The subject has an estimated life expectancy of more than 5 years
* The subject has confirmed stress urinary incontinence (SUI) through medical history, urodynamics, and/or physical exam for at least 6 months
* The subject has intrinsic sphincter deficiency due to one of the following:

post-TURP, simple open prostatectomy, radical prostatectomy completed at least 6 months prior to implantation date

* Positive Cough Stress Test (CST):
* Positive 24-hours Pad Test (PT):

A positive PT is confirmed with leakage of >8.O g/24h and < 400 g

* The subject has completed urodynamics, uroflow, post-void residual, and cystoscopy as per the protocol within 6 months prior to implant
* The subject is able and willing to complete all follow-up visits and procedures indicated in this protocol
* The subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the local ethics commit-tee of the respective site

Exclusion Criteria:

* Subjects who meet any of the following criteria are excluded from entry into the study
* The subject is unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with all follow-up requirements according to the study protocol
* The subject has an active urogenital infection or active skin infection in region of surgery
* The subject has serious bleeding disorders
* The subject has incontinence due to neurogenic causes defined as multiple sclerosis, spinal cord/brain injury, CVA, detrusor-external sphincter dyssynergia, Parkinson's disease, or similar conditions
* The subject had a previous implant to treat stress urinary incontinence
* The subject has undergone radiation, cryosurgery, or brachy therapy to treat prostate or other pelvic cancer within 6 months
* The subject is likely to undergo radiation therapy within the next 6 months
* The subject has active urethral or bladder neck stricture disease, requiring continued treatment
* The subject has urge predominant incontinence
* The subject has an atonic bladder or a postvoid residual (PVR) ≥150mL
* The subject has a condition or disorder likely to require future transurethral procedure
* The subject is enrolled in a concurrent clinical trial of any treatment (drug or device) that could affect continence function without the sponsors'approval
* Subjects who in the opinion of the investigator are unable and/or unlikely to to comprehend the nature, scope and possible consequences of the study and to follow the study procedures and instructions and complete all study related measurements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction using the Patient Global Impression of Improvement (PGI-I) score and assess change in 24-hour pad weight . | 12 months

SECONDARY OUTCOMES:
Assess change in subject satisfaction using questionnaires: ICIQ, UCLA-RAND Incontinence Index. | 12 months

OTHER OUTCOMES:
Summarize all cumulative device and procedure related adverse events | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada